CLINICAL TRIAL: NCT04509856
Title: The Impact Of Teach-Back Educational Method On Diabetes Knowledge Level And Clinical Parameters In Type 2 Diabetes Patients Undergoing Insulin Therapy
Brief Title: Teach-Back Educational Method On Diabetes Knowledge Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Yasemin Cayir, Clinical Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YaseminC
Record Dates: First submitted 2020-08-07; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Patient Empowerment
Keywords: diabetes; education; teach-back
MeSH Terms: conditions — Patient Participation; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Routine diabetes education will given to the patients included in the Control Group by a diabetes education nurse. The diabetes education nurse has been working for 10 years in the same center.
- Intervention Group (Experimental): Intervention Group will take their diabetes education by teach-back educational strategy.
  Interventions: Behavioral: Teach-back educational method

INTERVENTIONS:
Behavioral: Teach-back educational method — In the teach-back method, after teaching new information to the patient, the patients were asked to explain that new information in their own words. Then the patients' knowledge and the adequateness of their explanations were determined. The patient should repeat the instructions in their own words. In this way, the healthcare professional can evaluate how the patient understands the information. If the patient repeated the information correctly, the teach-back phase for that information was completed, and progression for new information was resumed. However, if there was a deficiency or error in the information, it was corrected and repeated by the healthcare professional.
  Arms: Intervention Group

SUMMARY:
It was aimed to research the effect of teach-back educational method on diabetes knowledge level and clinical parameters in type 2 diabetes patients undergoing insulin therapy. This is a randomized-controlled trial. Teach-back method will used for intervention group, routin diabetes education will used for control group. The primary outcome is diabetes knowledge levels (DKL), and secondary outcome is clinical patameters (fasting blood glucose, HbA1c, blood pressure). DKL and clinical parameters will measured and compared between two groups before and three months after the interventions.

ELIGIBILITY:
Inclusion Criteria:

* To have Type 2 Diabetes
* To be over 18 years old
* Not have any barriers in understanding and speaking Turkish
* Who started insulin treatment for the first time

Exclusion Criteria:

* Patients with a diagnosis of dementia
* To have vision or hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Diabetes knowledge level (DKL) | 3 months
  The DKL will be measured through a self-structured questionnaire containing 11 items. The questionnaire contains three answers: "yes," "no," or "I do not know." The right answer will be accepted as two points, the wrong answer as zero points, and the "I do not know" answer will be accepted as one point. The total scores ranges from 0-22. Higher scores of the questionnaire indicates that the higher DKL.

SECONDARY OUTCOMES:
Fasting blood glucose | 3 months
  Fasting blood glucose in mg/dl
HbA1c | 3 months
  HbA1c in %
Blood pressure | 3 months
  Blood pressure in mmHG

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Cayir, 1, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University Hospital, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The clinical outcomes will be shared.